CLINICAL TRIAL: NCT02622711
Title: Promoting Weight Loss Through Diet and Exercise in Overweight Women With Breast Cancer: A Four-arm Randomized Trial
Brief Title: Promoting Weight Loss Through Diet and Exercise in Overweight Women With Breast Cancer
Acronym: InForma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: European Institute of Oncology (Other)
Collaborators: Associazione Italiana per la Ricerca sul Cancro (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IEO 0244
Record Dates: First submitted 2015-11-06; First posted 2015-12-04 (Estimated); Last update posted 2020-01-30 (Actual); Status verified 2020-01

CONDITIONS: Breast Cancer
Keywords: breast cancer; obesity; weight control; exercise and physical fitness
MeSH Terms: conditions — Breast Neoplasms; Obesity; Motor Activity | interventions — Diet Therapy; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- DI Dietary Intervention (Experimental): Individualized dietary counselling to reduce body weight
  Interventions: Behavioral: DI
- PAI Physical Activity Intervention (Experimental): Individualized physical activity counseling to reduce body weight
  Interventions: Behavioral: PAI
- PADI Physical Activity+Diet Intervention (Experimental): Individualized dietary and physical activity counseling to reduce body weight
  Interventions: Behavioral: PADI
- LII Less Intensive Intervention (Experimental): Materials and guidelines available to general public
  Interventions: Behavioral: LII

INTERVENTIONS:
Behavioral: DI — Participants will be offered an individualized dietary counselling according to their lifestyle habits to reduce weight consisting of face-to face contacts, group meetings, motivational phone calls and information pamphlets.
  Other Names: Dietary Intervention
  Arms: DI Dietary Intervention
Behavioral: PAI — Participants will be offered an individualized physical activity counseling according to their lifestyle habits to reduce weight consisting of face-to face contacts, group meetings, motivational phone calls and information pamphlets.
  Other Names: Physical Activity Intervention
  Arms: PAI Physical Activity Intervention
Behavioral: PADI — Participants will be offered an individualized dietary and physical activity counseling to reduce weight consisting of face-to face contacts, group meetings, motivational phone calls and information pamphlets.
  Other Names: Physical Activity and Dietary Intervention
  Arms: PADI Physical Activity+Diet Intervention
Behavioral: LII — Participants will be considered as control group. They will receive a general healthy counselling providing materials and guidelines available for the general public.
  Other Names: Less Intensive Intervention
  Arms: LII Less Intensive Intervention

SUMMARY:
The investigators aim to evaluate the effect of a 6-month intervention (counseling) focused on weight loss in a group of overweight or obese women previously treated for early breast cancer. Intervention is designed to improve adherence to a healthy diet or/and to increase physical activity and decrease sedentary time, taking advantage of a pedometer-like device.

DETAILED DESCRIPTION:
The InForma project is designed as a mono-institutional randomized controlled 4-arm parallel-group trial. Potential study participants will be recruited among all overweight or obese breast cancer patients previously treated at the European Institute of Oncology (IEO). Potential study participants will be recruited after breast cancer treatments (surgery, chemotherapy and and/or radiation) will be completed. Study participants will be randomized to one of the 4 arms: DI - Dietary Intervention; PAI - Physical Activity Intervention; PADI - Physical Activity and Dietary Intervention; LII - Less Intensive Intervention. Enrolled patients will receive a 6-month intervention and will be followed until the end of the study period with two additional follow-up visits at 12- and 24-month. The main aim of the study is to evaluate the impact of the intervention programme on body weight change in overweight or obese breast cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with a first invasive non-metastatic breast carcinoma histologically confirmed,
* BMI > 25,
* within 6-month/one year of completion of main cancer treatment,
* being able to participate in the intervention,
* agree to wear the wrist-based activity monitor during the study period,
* agree to be randomized to either group,
* written informed consent.

Exclusion Criteria:

* severe medical condition or advanced age impeding the patient to adhere at the planned study follow-up period,
* contraindications to exercise due to history of heart condition, stroke, chest pain during activity or rest, severe hypertension
* orthopaedic disability that would prevent optimal participation in the physical activities prescribed,
* patient is unable to find transportation to the study location over the study period, - or
* plans to move away from Lombardy or to be out of town for more than 3 weeks during the study period.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 262 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Body weight reduction | baseline - 6 month
  weight loss ≥5% of the baseline body weight via calibrated scales, stadiometer

SECONDARY OUTCOMES:
Long-term body weight control | baseline - 12 month - 24 month
  long-term weight control or maintenance via calibrated scales, stadiometer
Pedometer Step Count | baseline - 6 month - 12 month - 24 month
  change in total step count via pedometer device with electronic data transmission
Physical activity level | baseline - 6 month - 12 month - 24 month
  change in physical activity and inactivity levels via IPAQ-International physical activity questionnaire
Dietary intake | baseline - 6 month - 24 month
  change in dietary intake via Food Frequency Questionnaire
Quality of life | baseline - 6 month - 12 month - 24 month
  change in quality of life via Functional Assessment of Cancer Therapy-Breast (FACT-B)
Mood | baseline - 6 month - 12 month - 24 month
  change in mood via State-Trait Anxiety Inventory (STAI) questionnaires
Lipid Marker Change | baseline - 6 month - 24 month
  change in LDL, HDL, triglycerides and cholesterol assessed by blood samples
Oestradiol level | baseline - 6 month - 24 month
  change in oestradiol assessed by blood samples
Insulin level | baseline - 6 month - 24 month
  change in insulin assessed by blood samples
Glucose level | baseline - 6 month - 24 month
  change in glucose assessed by blood samples
C-reactive protein level | baseline - 6 month - 24 month
  change in C-reactive protein assessed by blood samples

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Maisonneuve, Principal Investigator — European Institue of Oncology
Locations (1):
- IEO Istituto Europeo di Oncologia, Milan, Italy

REFERENCES:
- [Derived] Gnagnarella P, Carioni G, Draga D, Raja S, Baggi F, Simoncini MC, Mazzocco K, Masiero M, Bassi FD, Peradze N, Zorzino L, Pravettoni G, Sieri S, Maisonneuve P. Dietary patterns and change in food consumption in overweight or obese breast cancer survivors: the InForma randomized intervention trial. Nutr Metab Cardiovasc Dis. 2026 Feb;36(2):104378. doi: 10.1016/j.numecd.2025.104378. Epub 2025 Oct 16. PMID 41145327
- [Derived] Gnagnarella P, Draga D, Baggi F, Simoncini MC, Sabbatini A, Mazzocco K, Bassi FD, Pravettoni G, Maisonneuve P. Promoting weight loss through diet and exercise in overweight or obese breast cancer survivors (InForma): study protocol for a randomized controlled trial. Trials. 2016 Jul 28;17:363. doi: 10.1186/s13063-016-1487-x. PMID 27464488